CLINICAL TRIAL: NCT03960073
Title: Chronic Kidney Disease and Heart Failure With Preserved Ejection Fraction: The Role of Mitochondrial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HM20015440
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Renal Insufficiency, Chronic; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Experimental): 20mg daily oral dose of MitoQ
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): Oral TTP placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — 4 week 20mg oral daily dose of Mito Q
  Arms: MitoQ
Dietary Supplement: Placebo — 4 week oral daily dose of TTP placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the role of mitochondrial derived oxidative stress on exercise capacity and arterial hemodynamics in HFpEF patients with and without chronic kidney disease.

DETAILED DESCRIPTION:
Heart failure is a public health epidemic affecting 6.5 million Americans. Heart failure with preserved ejection fraction (HFpEF) accounts for a large burden of heart failure with the incidence and cost associated with the disease projected to double in the next 20 years. The pathophysiology of HFpEF has not yet been fully elucidated and no proven therapies for improving outcomes in HFpEF currently exist, posing major diagnostic and therapeutic challenges. The addition of chronic kidney disease (CKD) presents a complicated cardio renal syndrome that manifests a distinctly different phenotype and exacerbates the diagnostic and therapeutic challenges of HFpEF. This study aims to address the urgent need to establish treatment targets and therapies by investigating potential underlying biological contributors to HFpEF and its symptoms.

Mitochondrial dysfunction is consistently reported in CKD and heart failure. Mitochondrial dysfunction has been implicated in cardiac, skeletal muscle and vascular dysfunction and is therefore an attractive target for a 'whole systems' therapeutic approach that would encompass exercise intolerance and abnormal blood vessel hemodynamics. A known contributor to and subsequent cyclical result of mitochondrial dysfunction is an abnormally heightened production of mitochondria derived oxidative stress. This study will address the role of mitochondria derived oxidative stress in mitochondrial dysfunction, exercise intolerance and large blood vessel hemodynamics HFpEF patients with and without CKD.

ELIGIBILITY:
Inclusion Criteria:

1. above the age of 18 years
2. a clinical diagnosis of stable Stage C Heart Failure with NYHA Class II-III symptoms
3. a left ventricular ejection fraction >50%

Exclusion Criteria:

1. current cancer
2. current pregnancy
3. current antioxidant supplement use and unwilling to have a 7-day antioxidant washout period before the beginning the trial and to continue antioxidant disuse throughout the trial.
4. current antiretroviral medication use
5. absolute contraindications to exercise testing according to the American College of Sports Medicine guidelines
6. fluid overload
7. unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Change over 4 weeks
  Maximal aerobic capacity (VO2peak) obtained from cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Reflected Pulse Wave Amplitude | Change over 4 weeks
  Late systolic pulsatile load on the left ventricle represented by reflected pulse wave amplitude; assessed by echocardiography combined with applanation tonometry.
Forward Pulse Wave Amplitude | Change over 4 weeks
  Central hemodynamic assessment of the forward pulse wave amplitude assessed by echocardiography combined with applanation tonometry.
Mitochondrial Respiration | Change over 4 weeks
  High resolution mitochondrial respirometry

CONTACTS AND LOCATIONS:
Overall Officials: Danielle L Kirkman, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No